CLINICAL TRIAL: NCT00004856
Title: A Phase II Trial of Trastuzumab (Herceptin; NSC #688097, IND #6667) in Patients With Previously Treated Advanced Urothelial Tract Transitional Cell Carcinoma
Brief Title: Trastuzumab in Treating Patients With Previously Treated, Locally Advanced, or Metastatic Cancer of the Urothelium
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02046; CALGB 90101; UCSF-99535; CALGB-90101; CDR0000067476; NCI-T99-0108; U10CA031946 (NIH)
Record Dates: First submitted 2000-03-07; First posted 2003-09-30 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Distal Urethral Cancer; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Proximal Urethral Cancer; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment: Herceptin (Experimental): Patients receive a loading dose of trastuzumab (Herceptin) IV over 90 minutes on day 1 of week 1. For all subsequent doses, patients receive trastuzumab IV over 30 minutes weekly. Treatment may continue for more than 1 year in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: trastuzumab

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2

SUMMARY:
Phase II trial to study the effectiveness of trastuzumab in treating patients who have previously treated, locally advanced, or metastatic cancer of the urothelium. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate in patients with previously treated, locally advanced or metastatic transitional cell carcinoma of the urothelium treated with trastuzumab (Herceptin).

II. Determine the safety of this drug in this patient population. III. Determine overall and progression-free survival of this patient population treated with this drug.

OUTLINE:

Patients receive a loading dose of trastuzumab (Herceptin) IV over 90 minutes on day 1 of week 1. For all subsequent doses, patients receive trastuzumab IV over 30 minutes weekly. Treatment may continue for more than 1 year in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transitional cell carcinoma (TCC) of the urothelium, including the bladder, urethra, ureter, or renal pelvis

  * No pure adenocarcinomas, pure squamous cell carcinomas, small cell carcinoma, or only small foci of TCC (less than 10% of tumor specimen)
  * Locally advanced (T4b) TCC of the bladder
  * Metastatic (N2 or N3 or M1)TCC of the urothelium
  * HER2 expression (3+) as determined by immunohistochemistry or gene amplification by fluorescent in situ hybridization
* Must not be a candidate for potentially curative surgery or radiotherapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion of at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following lesions are considered nonmeasurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Primary bladder masses
* Relapsed from or failed to achieve a complete or partial response after 1 prior systemic chemotherapy regimen for TCC, including cisplatin, carboplatin, paclitaxel, docetaxel, or gemcitabine

  * Prior adjuvant or neoadjuvant chemotherapy is considered 1 prior chemotherapy regimen
  * Prior single-agent chemotherapy as a radiosensitizer is not considered a prior systemic chemotherapy regimen
* No known brain metastases
* Performance status - CTC 0-2
* More than 12 weeks
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 2 times ULN
* Creatinine clearance at least 30 mL/min
* Ejection fraction at least 50% (or lower limit of normal) by echocardiogram or MUGA
* No history of ongoing congestive heart failure
* No active cardiac ischemia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* HIV negative
* No known autoimmune disease
* No prior trastuzumab (Herceptin)
* At least 14 days since prior radiotherapy
* At least 30 days since prior chemotherapy
* Prior doxorubicin allowed provided cumulative dose is no greater than 300 mg/m^2
* Prior epirubicin allowed provided cumulative dose is no greater than 600 mg/m^2
* No concurrent chemotherapy
* No concurrent hormonal therapy except:

  * Steroids given for adrenal failure
  * Hormones administered for nondisease-related conditions (e.g., insulin for diabetes)
  * Intermittent dexamethasone as an antiemetic or for sensitivity reactions to study drug
* No concurrent palliative radiotherapy
* Prior radiotherapy allowed provided treated area is not only site of measurable disease
* At least 14 days since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-07; Primary Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete or partial response) as assessed by RECIST criteria | 1 year

SECONDARY OUTCOMES:
Toxicities as graded according to the NCI Common Toxicity Criteria | 12 weeks
Proportion of patients who are HER2 positive (3+ by IHC or FISH positive) | Baseline
Overall survival (OS) | From date of initiation of treatment to date of death due to any cause, assessed up to 1 year
Disease-free survival (DFS) | From date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arif Hussain, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States